CLINICAL TRIAL: NCT06319352
Title: Evaluation of Quality-of-Life Improvements Using UroShield for Patients Living in Long Term Care Facilities With Indwelling Urinary Catheters - A Pilot Study
Brief Title: Evaluation of Quality-of-Life Improvements Using UroShield Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Nanovibronix (Industry)
Responsible Party: Principal Investigator, Lona Mody, Principal Investigator, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: HUM00243293
Record Dates: First submitted 2024-03-12; First posted 2024-03-20 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Quality of Life; Catheter-Associated Urinary Tract Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active UroShield (Experimental): Active UroShield Device
  Interventions: Device: Active UroShield
- Sham UroShield (Sham Comparator): Inactive UroShield device
  Interventions: Device: Sham UroShield

INTERVENTIONS:
Device: Active UroShield — Participants will have an active device (i.e., ultrasound energy is being produced by actuator) attached to their urinary catheter tube.
  Arms: Active UroShield
Device: Sham UroShield — Participants will have an inactive device (i.e., no ultrasound energy being produced by the actuator) attached to their urinary catheter tube. All other aspects of the sham device (look, weight, feel, sound, and operation) are identical to the active device.
  Arms: Sham UroShield

SUMMARY:
The goal of this pilot study is to test key elements of the full study that will follow, including recruitment and retention strategies, intervention delivery, laboratory testing, data collection methods, and adherence to study protocol.

The main questions the investigators aim to answer focus on implementation and practicality:

* Recruitment feasibility and time to recruit
* How well do participants adhere to device protocol?
* How often do device components (i.e., actuators and drivers) have to be replaced?
* How much time is required for data collection and what sources or methods for data collection are used?

Results of this pilot study will inform the investigators as to necessary protocol modifications and overall feasibility for the larger randomized clinical trial to follow.

DETAILED DESCRIPTION:
The UroShield® device works by generating ultrasonic waves to interfere with attachment of bacteria inside the catheter, preventing biofilm formation and subsequent infections.

This double-blind pilot study aims to recruit 10-20 patients with urinary catheters (urethral or suprapubic catheters) living in nursing homes (NHs) in Michigan. Patients who consent to participate in the study will be randomized to either the treatment or control group and will have either an active treatment UroShield® device attached or a sham UroShield® device attached to the external tubing of their urinary catheter. Participants will wear the device continuously for a maximum of 90 days. Assessments of pain and quality-of-life will be conducted by study staff over a maximum of 6 study visits, along with clinical data collection via medical record review. A urine sample and catheter sample will also be collected by study staff at each catheter change (approximately every 30 days).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18+
* Indwelling urinary catheter (urethral or suprapubic) in place
* Written informed consent (and assent, when applicable) obtained from participant or participant's legal representative
* Able to comply with the requirements of the study

Exclusion Criteria:

* Pregnant or breastfeeding women
* Antibiotic use in past 10 days
* Ineligible catheter type in place (e.g., antimicrobial coated, 3-way catheter, condom catheter, nephrostomy tube, wicking device)
* Participation in another drug or device study in past 30 days
* History of poor compliance to medical treatment regimens
* Conditions that may severely compromise their ability to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Summarized every month for 6 months, or until the recruitment goal is reached.
  Number of patients enrolled out of number of patients eligible to participate in the study.

SECONDARY OUTCOMES:
Device use adherence | Summarized every month for at least 6 months, or until the recruitment goal is reached.
  Number of patients with at least 80% adherence out of total patients enrolled. Device adherence will be assessed via direct observation by study staff as well as patient/caregiver/clinician-reported (via written documentation or phone/email correspondence).
Device accountability | Summarized every month for at least 6 months, or until the recruitment goal is reached.
  Number of devices used out of the number of devices received. Extra components of the device (i.e., actuators) will be available to the study team; monitoring their use will validate amount and type of resources needed for intervention implementation.
Efficiency of data collection | Summarized every month for at least 6 months, or until the recruitment goal is reached.
  Time required for survey completion and data abstraction via chart review (actual time/expected time).

CONTACTS AND LOCATIONS:
Overall Officials: Lona Mody, Principal Investigator — University of Michigan
Locations (1):
- Evangelical Home - Saline, Saline, Michigan, United States